CLINICAL TRIAL: NCT03207373
Title: Reproducibility and Validity of the Stress ECG Test for the Evaluation of the Risk of Sudden Cardiac Death in a Paediatric Cohort With Preexcitation (WPW Pattern)
Brief Title: Stress ECG Test for the Evaluation of the Risk of Sudden Cardiac Death in a Paediatric Cohort With WPW Pattern
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study aim was not relevant anymore because other studies became available recently on the same topic
Sponsor: Christian Balmer (Other)
Responsible Party: Sponsor-Investigator, Christian Balmer, Head of Electrophysiology, principal investigator, clinical lecturer, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016-01943
Record Dates: First submitted 2017-03-08; First posted 2017-07-02 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Wolff-Parkinson-White Syndrome; Sudden Cardiac Death; Risk Stratification
MeSH Terms: conditions — Wolff-Parkinson-White Syndrome; Death, Sudden, Cardiac | interventions — Exercise Test; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stress ECG Test (Experimental): The whole study cohort undergoes the same diagnostic workup including stress test (ECG)
  Interventions: Diagnostic Test: Stress test (ECG)

INTERVENTIONS:
Diagnostic Test: Stress test (ECG) — Every study participant undergoes a standard diagnostic stress ECG

SUMMARY:
Patients with preexcitation are at risk for sudden cardiac death. The pathogenesis is a rapid antegrade conduction of atrial fibrillation over the accessory pathway to the ventricle resulting in ventricular fibrillation. Today it is possible to eliminate the conduction over the accessory pathway by catheter intervention (radiofrequency ablation) with a low rate of complications and a high rate of success. In clinical practice it is therefore important to estimate the risk for sudden cardiac death in an individual patient to give an advice to the patient and the parents about the further evaluation and therapeutic strategy. The velocity of the conduction over the accessory pathway can be estimated by analysing the ECG during sinus tachycardia. If the preexcitation disappears at a relatively low heart rate, the risk for sudden death is less than in patients with persisting preexcitation at the maximal heart rate. Compared to the gold standard i.e. measurement of the refractory period of the accessory pathway during invasive electrophysiological study (EPS), the measurements at the stress ECG have been reported to be a relatively poor indicator for an elevated risk which may be explained by a high intraindividual variability of this test. This study is designed to define the clinical relevance of the stress ECG in paediatric patients with preexcitation (compared to the invasive electrophysiological study).

First Hypothesis:

The results of the 3 stress ECG-tests are reproducible in an individual patient.

Null hypothesis: there is no difference between the three measurements of cycle length during stress ECG. Alternate hypothesis: the difference between the three measurements of cycle length is > 10%.

Second Hypothesis:

There is a close correlation between the results at stress ECG and the results at the invasive electrophysiological Intervention.

DETAILED DESCRIPTION:
Single centre, interventional study. There will be no randomisation or blinding.

This study evaluates the stress ECG test as a non-invasive method of risk stratification in patients with WPW syndrome. For the non-invasive part a stress electrocardiogram on a treadmill is used. The invasive comparison is made with an electrophysiological study (EPS) in the catheterization laboratory. Nowadays the gold standard for measuring the antegrade effective refractory period of the accessory pathway is the invasive EPS.

Study category A; there is only a minimal risk and a minimal burden to the study participants; The stress ECG test is a recommended test for this specific patient group as indicated in international guidelines.

The responsible investigator at the single study site ensures that approval from an appropriately constituted Competent Ethics Committee (CEC), is sought for the clinical study.

Objectives: 1) The study seeks primarily to evaluate the reproducibility of the loss of the preexcitation in repetitive stress ECG test in paediatric patients with WPW pattern in the view of an accurate estimation of the individual risk for sudden cardiac death.

2) To compare the results of non-invasive ECG measurements with measurements taken during invasive EPS and clinical/anatomical parameters.

Planned Analysis: Descriptive statistic is applied to all clinical parameters. All the 3 cycle lengths out of the stress ECG are compared individually with the ERP-AP from the invasive EPS. If there is an average from the cycle length, this would be compared with the ERP-AP as well. And then we compare whether the difference between the cycle length and the ERP-AP is similar in a group of patients (high/low risk) or even in all patients.

To demonstrate those results we use the Bland-Altman plot. There will also be a graph with the distribution of age of all patients. It will be interesting to see whether the age influences the results for example in relation to high or low risk.

After the EPS, the patients are divided into 2 risk categories: high risk (ERP-AP ≤ 250 ms) and low risk (ERP-AP > 250ms) as measured at the EPS.

At the end a risk factor analysis is made. All the parameters out of the case report form will be analysed whether the patient has high or low risk.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Preexcitation in resting ECG (WPW ECG Pattern)
* Age between 8 and 18 years
* Invasive EPS must be indicated/planned at the Children's Hospital Zurich

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems or psychological disorders of the participant
* Inability to walk/run on a treadmill

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Cycle length (CL) at the Stress ECG Test | 3 test within a month
  Cycle length (ms) at the point when the delta wave disappears and/or at the point of maximal heart rate (HR) (ms)

SECONDARY OUTCOMES:
ERP-AP from invasive EPS | 1 single measurement at aprox 1 month
  Effective Refractory Period of Accessory Pathways (ERP-AP) during programmed atrial pacing (ms)
SPERRI from invasive EPS | 1 single measurement at aprox 1 month
  Shortest pre excited Interval between two cardiac cycles (SPERRI)
Anatomical localisation of the AP measured in the EPS | 1 single measurement at aprox 1 month
  leftsided (superior, posterosuperior, posterior, posteroinferior, inferior) or rightsided (paraseptal, inferior, anteroinferior, anterior, anterosuperior and superior)

OTHER OUTCOMES:
Heart rate of 12-lead Resting ECG | 1 single measurement within 1 month
  (bpm)
Rhythm during 12-lead Resting ECG | 1 single measurement within 1 month
  sinus rhythm yes/no
axis of the QRS complex out of the 12-lead Resting ECG | 1 single measurement within 1 month
  (degree)
Duration of PQ Interval out of the 12-lead Resting ECG | 1 single measurement within 1 month
  (ms)
Duration of the QRS complex (ms) out of the 12-lead Resting ECG | 1 single measurement within 1 month
  (ms)
Z-value of left ventricle (LV) out of Echocardiography | 1 single measurement at aprox 1 month
  Z-value LV
Z-value of right ventricle (RV) out of Echocardiography | 1 single measurement within 1 month
  Z-value RV
Z-value of left Atrium (LA) out of Echocardiography | 1 single measurement within 1 month
  Z-value LA
Shortening fraction (SF) measured in Echocardiography | 1 single measurement within 1 month
  SF (%)
Ejection fraction (EF) measured in Echocardiography 5 | 1 single measurement within 1 month
  EF (%)
Valvular insufficiency measured in Echocardiography | 1 single measurement within 1 month
  aorta-, pulmonal-, tricuspidal-, mitral insufficiency (no, minimal, moderate, severe)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Balmer, PD Dr. med., Principal Investigator — University Childrens Hospital
Locations (1):
- University Childrens Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No